CLINICAL TRIAL: NCT04365647
Title: Intra-operative Variation in Size of Brain Tumors After Craniotomy - Observational Comparative Imaging Study
Brief Title: Intra-operative Variation in Size of Brain Tumors After Craniotomy
Status: Completed | Type: Observational
Sponsor: Sheri Kashmir Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Kaushal Deep Singh, Doctor, Sheri Kashmir Institute of Medical Sciences
Other Study IDs: SKIMS, Soura
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Brain Tumor, Primary
Keywords: Parenchymal brain tumors; Intraaxial brain tumors; Gliomas; Glioblastoma multiforme; Low grade glioma; High grade glioma; Intraoperative Ultrasound (IOUS); Tumor Surfacing; Tumor expansion; Contrast enhanced magnetic resonance imaging (CEMRI) brain; Contrast enhanced computed tomography (CECT) brain
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patient's in whom there is increase in tumor size after craniotomy
- 2: Patient's in whom there was either no increase in tumor size or decrease in tumor size after craniotomy

SUMMARY:
We planned to evaluate the change in tumor dimensions of intraaxial parenchymal tumors after craniotomy by comparing the tumor size on intraoperative ultrasonography (IOUSG) with pre-operative CECT and CEMRI brain.

DETAILED DESCRIPTION:
Background: No previous study to determine the intraoperative changes in the tumor dimensions had been undertaken previously. Objectives: We planned to evaluate the change in tumor dimensions of intraaxial parenchymal tumors after craniotomy by comparing the tumor size on intraoperative ultrasonography (IOUSG) with pre-operative CECT and CEMRI brain. Study Design: This was a prospective observational study. Participants: Patients aged 15-65 years undergoing surgery at SKIMS for intraaxial parenchymal intracranial tumors were included. Methods: Standard pre-operative CECT and CEMRI brain were done to measure tumor dimensions and compared with IOUSG.

ELIGIBILITY:
Inclusion Criteria:

* All patients above the age of 15 years conferring to Grade I and II of American Society of Anesthesiologist (ASA) physical status classification system, undergoing elective craniotomy with intracranial tumor excision were included in this study. Patients with or without any neuro-deficit were also included. Only those patients in whom all the tumor dimensions could be defined with precision on pre-operative CECT, CEMRI and IOUSG were included in the final analysis.

Exclusion Criteria:

* Patients' in whom there are multiple intracranial tumors (e.g. metastasis), deep seated tumors, inability to use IOUSG and in whom exact tumor dimensions cannot be defined either on pre-operative CECT/CEMRI or on IOUSG were excluded.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients above the age of 15 years conferring to Grade I and II of American Society of Anesthesiologist (ASA) physical status classification system undergoing elective intracranial tumor surgery at our institute in the specified period.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Tumor dimension change | March 2018 to November 2019
  Change in tumor dimension, surface area and volume when comparing intraoperative ultrasound with pre-operative CEMRI and CECT brain

SECONDARY OUTCOMES:
Tumor distance from dural surface | March 2018 to November 2019
  Change in the distance of tumor from dural surface as measured on intraoperative ultrasound when comparing it with pre-operative CEMRI and CECT brain
Relationship of tumor size change with other characteristics | March 2018 to November 2019
  Relationship of tumor size change with tumor consistency, tumor characteristics, histopathology, tumor location

CONTACTS AND LOCATIONS:
Overall Officials: Abdul R Bhat, MCh, Principal Investigator — Sher-i-Kashmir Institute of Medical Sciences, Soura
Locations (1):
- Sher-i-Kashmir Institute of Medical Sciences, Soura, Srinagar, Jammu and Kashmir, India

IPD SHARING:
Plan to Share IPD: No